CLINICAL TRIAL: NCT02961478
Title: Measurement of Iohexol Plasma Clearance in Patients Leaving ICU After Acute Renal Failure
Acronym: IOXSOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC2015-06
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iohexol plasmatic clearance (Experimental)
  Interventions: Drug: IOHEXOL

INTERVENTIONS:
Drug: IOHEXOL — Estimate iohexol clearance at the end of stay in intensive care for patients who had an episode of acute renal failure.
  Other Names: Omnipaque ®

SUMMARY:
IOXSOR study's purpose to determine the frequency of non resolutive renal failure (estimated by the clearance of iohexol) at end of stay in ICU patients who have had acute renal failure episode.

ELIGIBILITY:
Inclusion Criteria:

* ICU stay > 7 days
* Having presented during the stay renal failure stage 2 or 3 Kidney Disease Improving Global Outcomes (KDIGO)
* Steady improvement of renal function before the ICU discharge :

  * Creatinine before ICU discharge <110 µmol / L for women, <130 µmol / L for men
  * No recourse to extra renal purification
  * Change in creatinine levels (ΔCréatinine) less than 20% over two measures spaced 24 hours within 48 hours preceding the discharge
* Expected discharge ICU within 48 hours :

  * Glasgow score > 13
  * Lack of mechanical ventilation except home Noninvasive Mechanical Ventilation (NiMV)
  * Lack of use of catecholamine
  * No contra-indication for discharge according to physician in charge of the patient
* Informed consent signed by the patient, where not possible by the person of trust or the family if present. Written consent by the patient will be obtained as soon as deemed possible.

Exclusion Criteria:

* Iohexol administration within 48 hours preceding the potential inclusion (imaging examination with X-ray contrast medium injection)
* Iohexol administration planned within 24 hours after potential inclusion in the study
* Known medical history of immediate allergic or delayed skin allergic reaction to injection of iodinated contrast material or any serious doubt on this medical history
* Patient receiving from extra renal purification during ICU discharge
* Chronic renal disease known (creatinine> 110 µmol / L for women,> 130 µmol / L for men) or creatinine clearance estimated less than 60 mL / min
* Pregnancy or breastfeeding women
* Patient under guardianship or safeguard justice known at the time of inclusion
* Patient limitation care
* Person not affiliated or not the beneficiary of a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with a clearance of iohexol < 60 ml/min/1m273 at the end of ICU hospitalisation. | 24 hours
  Iohexol clearance pharmacokinetics

SECONDARY OUTCOMES:
Correlation between non resolutive renal at the end of ICU (iohexol clearance < 60 ml/min/1m273) and creatinine clearance < 60 ml/min/1m273 at 6 month after ICU. discharge | Six month after ICU discharge
Number of risk factors associated with non resolutive among : Age Previous renal function Comorbidities Severity parameters of renal aggression Acute severity of parameters during the ICU hospitalisation | 24 hours
Correlation between serum creatinine derived measurements of Glomerular Filtratio Rate and iohexol clearance. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: François BELONCLE, CCU-AH, Principal Investigator — University Hospital, Angers
Locations (5):
- France (5):
  - University Hospital, Angers
  - Hospital center, Chartres
  - Hospital, Le Mans
  - University Hospital, Poitiers
  - University Hospital, Tours